CLINICAL TRIAL: NCT01401738
Title: Results of Shoulder Arthroscopic Surgery for Rotator Cuff, Biceps Tendon, Labrum and Capsule
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Tai-Yuan Chuang, Department of Traumatology, Wanfang Hospital
Other Study IDs: 100008
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Shoulder Arthroscopic Surgery
Keywords: Shoulder Arthroscopic Surgery

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a retrospective review of chart. Clinical results including range of motion, muscle power and scores will be recorded. Arthroscopic surgery of rotator cuff, labrum and capsule well be re-evaluated for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder lesions including capsule, biceps, rotator cuff which indicated for arthroscopic surgery

Exclusion Criteria:

* Open surgery for shoulder lesions
* Concomitant open and arthroscopic surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Shoulder Arthroscopic Surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2011-05; Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Yuan Chuang, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan